CLINICAL TRIAL: NCT03968354
Title: NASH and Type 2 Diabetes: Role of the Receptor Activator of Nuclear Factor-κB (RANK) and Its Ligand (RANKL)
Acronym: NADRANK-1
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: K171105J; 2018-A02468-47 (Other: APHP-DRCI)
Record Dates: First submitted 2019-05-14; First posted 2019-05-30 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Diabetes type2; NASH - Nonalcoholic Steatohepatitis; NAFLD
Keywords: NAFLD; NASH; Diabetes type2
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — One additional blood tube will be collected for DNA collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Steatosis group - Experimental1: Steatosis group
  Interventions: Biological: "Collection of additional blood tubes; Biobanking (plasma, liver tissue).
- NASH group without fibrosis - Experimental 2: NASH group without fibrosis
  Interventions: Biological: "Collection of additional blood tubes; Biobanking (plasma, liver tissue).
- Moderate fibrosis - Experimental 3: Moderate fibrosis
  Interventions: Biological: "Collection of additional blood tubes; Biobanking (plasma, liver tissue).
- Advanced fibrosis - Experimental 4: Advanced fibrosis
  Interventions: Biological: "Collection of additional blood tubes; Biobanking (plasma, liver tissue).
- Control group - Active Comparator: Control group
  Interventions: Biological: "Collection of additional blood tubes; Biobanking (plasma, liver tissue).

INTERVENTIONS:
Biological: "Collection of additional blood tubes; Biobanking (plasma, liver tissue). — * Preservation of liver tissue obtain by liver biopsy, constitution of a collection
  * Sampling of additional blood tubes for a biological collection (serum): Serum biomarker research and genetic research

SUMMARY:
Non-alcoholic fatty liver diseases (NAFLD) include several entities ranging from simple steatosis to hepatic fibrosis or cirrhosis. Steatosis, considered benign and the first stage of the disease, is characterized by the accumulation of triglycerides in the liver. It may in some cases progress to nonalcoholic steatohepatitis (NASH), which is characterized by the presence of a marked inflammation with or without fibrosis. NAFLD is the most common liver disease in the world and is particularly associated with type 2 diabetes (T2D) (80% in the diabetic population). While NASH is characterized by a higher prevalence of mortality from a cardiac and hepatic (cirrhosis and cancer) origin, therapeutic resources are almost non-existent.

RANK (receptor activator of NF-kB) and its ligand RANKL (a member of the TNFalpha family) have emerged in recent years as new players in bone pathophysiology. By binding to its receptor, RANKL induces a number of signaling pathway and in particular the NF-kB pathway (Nuclear factor-kB), a major player in inflammation. Recent literature shows that the role of RANK / RANKL is not confined to the bone but may be involved in the genesis of inflammation in other tissues. It has been shown recently that a high circulating level of RANKL was a risk factor predictor of T2DM. Furthermore, the invalidation of RANK specifically in hepatocytes protects from insulin resistance and hepatic steatosis induced by a high fat diet in mice.

The aim of our project is to provide a proof of concept that the RANKL / RANK system plays an important role in the pathogenesis of NAFLD and in the progression of this disease to NASH. The aim of our project is to provide a proof of concept that the RANKL / RANK system plays an important role in the pathogenesis of NAFLD and in the progression of this disease to NASH.

The investigator propose to study the RANKL / RANK expression in serum and liver biopsies of type 2 diabetic patients at different stages of NAFLD.

DETAILED DESCRIPTION:
Objectives:

To show that (i) expression of mRNA and proteins of the RANKL pathway (RANK, RANKL, OPG) in liver and (ii) serum concentration of RANKL/OPG proteins are correlated with the gravity of the NAFLD.

Study protocol:

Identify patients with different stages of NAFLD (mere steatosis, NASH, and moderate or advanced fibrosis) from the database of patients who have undergone liver biopsy in the hepatology department of the Pitié-Salpêtrière Hospital . From the hepatic tissue, the paraffin-embedded liver biopsies and the serum of these patients, study of the expression of mRNA (quantitative RtPCR) and proteins (immunohistochemistry, western blots) of the RANKL pathway (RANK, RANKL, OPG) in liver. In the serum of these patients, measure of concentration of RANKL and OPG proteins as described above.

Study Type: monocentric, observational, case-control, analytical study Study duration: 18 months (time for data collection, for cellular biological experimentations and for data analysis)

Patient Population:

5 groups of patients very well phenotyped and with liver biopsy (with at our disposal frozen liver tissue, paraffin-embedded liver tissue and serum for all the patients):

* 1) steatosis group (n=10)
* 2) NASH group without fibrosis (n=10)
* 3) moderate fibrosis (n=10)
* 4) advanced fibrosis (n=10)
* 5) healthy control group without liver disease (n=10) Comprehensive clinical and laboratory data were observed at the time of the liver biopsy and are available for all the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients adults with type 2 diabetes
2. Patients with one of the following criteria:

   * Steatosis, defined on biopsy as either steatosis alone (≥5% hepatocytes with fat) or steatosis without evidence of ballooning, with spotty lobular inflammation of grade 1 maximum (<2 foci/sox power field) and no fibrosis (Steatosis group) OR
   * Patients with NASH, defined on biopsy, as steatosis (≥5%) co-existing with hepatocellular ballooning and lobular necroinflammation, without fibrosis (NASH group) OR
   * Fibrosis on biopsy, where fibrosis will be defined as moderate if fibrosis is perisiunsoidal or periportal fibrosis (F1) or perisinusoidal and periportal/portal (F2) (Moderate fibrosis) OR
   * Fibrosis on biopsy, where fibrosis will be defined as advanced if there is bridging fibrosis (F3) or cirrhosis (F4) (Advanced fibrosis group) OR
   * Patients without NAFLD: control population. Patients for whom a biopsy was performed due to liver biological abnormalities but without NAFLD criteria on biopsy OR patients with abdominal surgery during which a liver biopsy was performed and without NAFLD criteria on biopsy. (Control group).
3. Patient affiliated to social security;
4. Signed informed consent.

Exclusion Criteria:

1. Patients with liver diseases other than NAFLD (drug-induced hepatotoxicity, chronic hepatitis B or C, genetic hemochromatosis, autoimmune hepatitis, primary biliary cirrhosis, primary sclerosing cholangitis, α1-antitrypsin deficiency, Wilson's disease, etc.)
2. Patients with daily alcohol consumption higher than 30 g/d (men) and 20 g/d (women)
3. Patients exposed to drugs that can induce secondary NAFLD (corticosteroids, amiodarone, tamoxifen)
4. Patient unable or unwilling to understand and sign an informed consent form.
5. Patient deprived of liberty or under legal protection measure
6. Weight ≤ 40 kg
7. Patients with hemoglobin < 7 g/dL or 9 g/dL if existence of respiratory or cardiac disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We will constitute 5 groups of patients very well phenotyped and with liver biopsy (with at our disposal frozen liver tissue, paraffin-embedded liver tissue and serum for all the patients):
  1. steatosis group (n=10);
  2. NASH group without fibrosis (n=10);
  3. moderate fibrosis (n=10);
  4. advanced fibrosis (n=10);
  5. Control group (n=10).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Measure of RANKL mRNA expression in the liver | Baseline
  Expression of RANKL mRNA in liver of patients with NASH or NAFLD with fibrosis comparatively to patients with mere steatosis.

SECONDARY OUTCOMES:
Serum concentrations of RANKL | Baseline
  Measure of Serum RANKL concentration in patients with NASH or NAFLD with fibrosis comparatively to patients with mere steatosis and in NAFLD patients comparatively to healthy controls.
Serum osteoprotegerin concentrations | Baseline
  Measure of serum osteoprotegerin concentrations in type 2 diabetic patients with NASH or NAFLD with fibrosis compared to type 2 diabetic patients with simple steatosis and in patients with type 2 diabetes with NAFLD compared to healthy controls.
HOMA-IR | Baseline
  Correlation between RANK and RANKL protein expression and insulin resistance and correlation between serum concentrations of RANKL / osteoprotegerin and insulin resistance in type 2 diabetic patients with NASH and NAFLD with fibrosis compared to type 2 diabetic patients with simple steatosis and in patients with type 2 diabetes with NAFLD compared to healthy controls
Measure of RANKL mRNA | Baseline
  Expression of RANKL mRNA and RANKL protein in liver tissue of NAFLD patients comparatively to healthy controls.
Measure of RANKL protein levels | Baseline
  Expression of RANKL protein in liver of patients with NASH or NAFLD with fibrosis comparatively to patients with mere steatosis.
Measure of RANK mRNA | Baseline
  Expression of RANK mRNA and protein in liver of patients with NASH or NAFLD with fibrosis comparatively to patients with mere steatosis and in liver tissue of NAFLD patients comparatively to healthy controls
Measure of RANK protein levels | Baseline
  Expression of RANK protein in liver of patients with NASH or NAFLD with fibrosis comparatively to patients with mere steatosis and in liver tissue of NAFLD patients comparatively to healthy controls.
RANK/RANKL genes polymorphisms | Baseline
  Association between RANK/RANKL gene polymorphisms and NAFLD development To highlight association between RANK/RANKL genes polymorphisms and NAFLD development.
NF-kB pathway in hepatocytes and Kupffer cells | Baseline
  Correlation of liver RANKL and RANK proteins expression with activation of NF-kB pathway in hepatocytes and Kupffer cells of patients with NASH or NAFLD with fibrosis comparatively to patients with mere steatosis and in NAFLD patients comparatively to healthy controls and correlation of serum RANKL and osteoprotegerin concentrations with activation of NF-kB pathway in hepatocytes and Kupffer cells in NAFLD patients comparatively to healthy controls and in NAFLD patients comparatively to patients with mere steatosis.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier MD, PHD Bourron, Principal Investigator — Hopital Universitaire La Pitié-Salpêtrière